CLINICAL TRIAL: NCT01554254
Title: Evaluation of the Safety and Efficacy of TXA127 (Angiotensin 1-7) to Enhance Engraftment in Pediatric Patients Undergoing Single or Double Umbilical Cord Blood Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Tarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXA127-2010-002
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Cord Blood Transplant; Hematologic Malignancy; Inherited Metabolic Disease
Keywords: Cord blood transplant; hematological malignancy; inherited metabolic disease; Mucositis; Neutrophil engraftment; Platelet recovery; Immune reconstitution
MeSH Terms: conditions — Hematologic Neoplasms; Mucositis | interventions — angiotensin I (1-7)

ARMS (1):
- 300mcg/kg/day for 28 days (Experimental)
  Interventions: Drug: TXA127

INTERVENTIONS:
Drug: TXA127 — 300mcg/kg/day, subcutaneous injection for up to 28 days

SUMMARY:
Engraftment failure is a major obstacle to the success of cord blood transplantation in children with malignancies and inherited metabolic disorders, despite the fact that they receive relatively high doses of nucleated cells from UCB. TXA127 is pharmaceutically formulated Angiotensin 1-7 [A(1-7)], a non-hypertensive derivative of Angiotensin-II (which contains the 8th amino acid conferring receptor binding to blood pressure receptors). TXA127 has multilineage effects on hematopoietic progenitors in vitro and in vivo. Preclinical data show that TXA127 is a novel stimulator of early multilineage hematopoietic progenitors, increases engraftment of committed hematopoietic progenitors, and induces more rapid production of platelets and neutrophils in the peripheral circulation, especially in limited cell number transplants. Treatment with TXA127 following UCBT is expected to increase the numbers of hematopoietic progenitors and accelerate engraftment.

ELIGIBILITY:
Inclusion Criteria:

* Subject, parent, or legal guardian provided written informed consent.
* Subjects must be >6 months and <21 years of age.
* Subjects must have one or two available 4, 5, or 6/6 antigen matching unrelated UCB unit(s) that will deliver a cell dose between 3.0-5.0 x 107cells/kg.

  * These units must be HLA-matched minimally at 4 of 6 HLA-A and B (at intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing) loci with the subject.
  * If two CB units will be used, the units must be HLA-matched at 3 of 6 HLA- A, B, and DRB1 loci with each other (using same resolution of molecular typing as indicated above).
  * For a single unit transplant, a minimum of 3 x 107cells/kg will be required.
  * For a double unit transplant, HLA-matched units must be available such that together both units deliver a combined pre-cryopreserved nucleated cell dose of at least 4.0 x 107 cells/kg with 1 unit of at least 2.5 x 107 cells/kg and the other at least 1.5 x 107 cells/kg.
* Subjects must have histologically confirmed diagnosis of a hematologic malignancy or a laboratory confirmed inherited metabolic disease.
* Subjects who have had a prior autologous or allogeneic transplant are allowed to participate provided it has been >1 year since the transplant was completed.
* Subjects must not have active CNS disease at the time of study enrollment.
* Subjects must have a life expectancy of >4 months.
* Female subjects capable of reproduction (defined as a subject who has started menses) must agree to the following:

  * Use of an effective oral or IM contraceptive method during the course of the study and 2 months following the last administration of study drug.
  * Female subjects capable of reproduction must have a negative pregnancy test result within 3 days prior to first study drug dose.
* Subjects must have adequate function of other organ systems as measured by:

  * Creatinine <2.0 mg/dL and creatinine clearance >50 mL/min.
  * Hepatic transaminases (ALT/AST) <4 x ULN, bilirubin <2.0 mg/dL.
  * Adequate cardiac function by echocardiogram or MUGA scan (ejection fraction or shortening fraction >80% of normal value for age).
  * Pulmonary function tests demonstrating FVC and FEV1 of >60% of predicted. DLCO should be used for subjects >10 years old. Crying vital capacity of >60% may be substituted for subjects unable to complete PFTs.

Exclusion Criteria:

* Subjects with an uncontrolled infection at the time of cytoreduction.
* Subjects who are pregnant or breast feeding.
* Subjects who are known to be seropositive for HIV or HTLV-1.
* Subjects who have had an autologous or allogeneic transplant <1 year from the anticipated administration of the first dose of study drug.
* Subjects who have received treatment with an investigational agent within 30 days of anticipated administration of the first dose of study drug.
* Subjects with current alcohol use, illicit drug use or any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the subject's ability to comply with the study requirements or visit schedule.
* Subjects must not have any co-morbid condition which, in the view of the Principal Investigators, renders the subject at too high a risk from treatment complications and regimen-related morbidity/mortality.

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety of TXA127 in subjects undergoing cord blood transplantation | Through Day 100 post transplant

SECONDARY OUTCOMES:
Effect of TXA127 on incidence, severity and duration of aGVHD | Through Day 100 post transplant
Effect of TXA127 on incidence, severity and duration of mucositis | Through Day 100 post transplant
  WHO oral toxicity score
Effect of TXA127 on neutrophil engraftment | Through Day 100 post transplant
Effect of TXA127 on platelet recovery | Through Day 100 post transplant
Effect of TXA127 on immune reconstitution | Through Day 100 post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Page, MD, Principal Investigator — Duke University; Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Pediatric Bone and Cord Blood, Duke Univ. Med. Center, Durham, North Carolina, United States